CLINICAL TRIAL: NCT05998941
Title: TQB2868 Plus Platinum-based Chemotherapy With or Without Bevacizumab in the First-line Treatment of Persistent, Recurrent, or Metastatic Cervical Cancer: a Single-arm, Open-label Phase Ⅱ Study
Brief Title: A Trial of TQB2868 Plus Platinum-based Chemotherapy With or Without Bevacizumab in the First-line Treatment of Persistent, Recurrent, or Metastatic Cervical Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow progress in development, the sponsor decided to withdraw and no longer proceed.
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2868-II-01
Record Dates: First submitted 2023-08-08; First posted 2023-08-21 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Paclitaxel; Cisplatin; Carboplatin; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2868 injection + Paclitaxel injection + Cisplatin/Carboplatin injection ± Bevacizumab injection (Experimental): TQB2868 injection + paclitaxel injection + cisplatin/carboplatin injection ± bevacizumab injection, 3 weeks (21 days) as a treatment cycle.
  Interventions: Drug: TQB2868 injection; Drug: Paclitaxel injection; Drug: Cisplatin injection; Drug: Carboplatin injection; Drug: Bevacizumab injection

INTERVENTIONS:
Drug: TQB2868 injection — TQB2868 injection is an anti-programmed cell death protein 1 (PD-1)/ transforming growth factor-β (TGF-β) dual-function fusion protein.
Drug: Paclitaxel injection — Paclitaxel injection prevents depolymerization of microtubules, inhibits mitosis, and hinders normal cell division.
Drug: Cisplatin injection — Cisplatin injection can inhibit the DNA replication process of cancer cells
Drug: Carboplatin injection — Carboplatin injection acts directly on DNA, thus inhibiting the vigorous division of tumor cells.
Drug: Bevacizumab injection — Bevacizumab is a humanized monoclonal antibody against vascular endothelial growth factor (VEGF).

SUMMARY:
This study used a single-arm, open phase II multicenter trial design. All eligible subjects received TQB2868 plus platinum-based chemotherapy with or without bevacizumab. A total of 39 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed persistent, recurrent or metastatic (International Federation of Gynecology and Obstetrics (FIGO) stage IVB) cervical cancer with squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma;
* It is not suitable for radical treatment such as surgery, radiotherapy and concurrent chemoradiotherapy;
* No previous systemic therapy for persistent, recurrent or metastatic cervical cancer;
* Provide archived or freshly obtained tumor tissue samples within the past 2 years or provide traceable test reports;
* 18 years old ≤75 years old (calculated on the date of signing the informed consent); Eastern Cooperative Oncology Group (ECOG) score 0-1; Expected survival ≥3 months;
* At least one measurable lesion according to (Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria;
* The main organs function well and meet the following standards:

  1. Blood routine test criteria (in the case of no blood transfusion and no correction by hematopoietic stimulating factor drugs within 14 days before screening) : absolute neutrophil count (ANC) ≥1.5×109 /L; Platelet ≥100×109 /L; Hemoglobin ≥100 g/L.
  2. Blood biochemical tests should meet the following criteria: total bilirubin (TBIL) ≤2× upper limit of normal (ULN) (≤3×ULN in Gilbert syndrome patients); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN. If liver metastasis is present, ALT and AST≤5×ULN; Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance ≥60 mL/min; Serum albumin (ALB) ≥30g/L.
  3. Urine routine examination criteria: urine routine indicated that urinary protein <++; If urinary protein ≥++, it should be confirmed that 24-hour urinary protein quantification ≤1.0 g.
  4. Coagulation function test criteria: prothrombin time (PT), activated partial thromboplastin time (APTT), international normalized ratio (INR) ≤1.5×ULN (no anticoagulant therapy).
  5. Thyroid stimulating hormone (TSH) ≤ ULN; If abnormal, T3 and T4 levels should be examined. If T3 and T4 levels are normal, they can be selected.
  6. Echocardiographic assessment: left ventricular ejection fraction (LVEF) ≥50%.
  7. 12-lead Electrocardiograph (ECG) assessment: Corrected QT interval prolongation (QTc)<470ms (female).
* Female subjects of childbearing age should agree to use contraception (such as intrauterine device (IUD), birth control pill or condom) during the study period and within 6 months after the study. A negative serum or urine pregnancy test within 7 days prior to study entry and must be non-lactating.
* Subjects voluntarily participated in this study, signed informed consent, and had good compliance.

Exclusion Criteria:

* Tumor disease and medical history:

  1. Have developed or are currently suffering from other malignant tumors within 3 years. The following two cases were included: other malignant tumors treated by single surgery, achieving R0 resection and no recurrence or metastasis; Cured non-melanoma skin cancer, nasopharyngeal carcinoma, and superficial bladder tumors
  2. Other pathological types, such as mucinous adenocarcinoma, clear cell adenocarcinoma, neuroendocrine tumor;
  3. tumor infiltration into the bladder or rectum;
  4. Subjects with known central nervous system (CNS) metastases and/or carcinomatous meningitis;
  5. Patients whose imaging showed that the tumor had invaded important blood vessels or the investigators judged that the tumor was highly likely to invade important blood vessels during the follow-up study and cause fatal hemorrhage;
  6. Uncontrollable pleural, pericardial, or peritoneal effusions requiring repeated drainage.
* Previous anti-tumor therapy:

  1. Received the last concurrent chemoradiotherapy for radical surgery or postoperative adjuvant therapy within 3 months before the first medication; Received palliative radiotherapy within 2 weeks before the first dose;
  2. Previously received platinum-based dual agents or any other chemotherapy agents in concurrent chemoradiotherapy for radical purposes;
  3. Received Chinese patent medicine with anti-tumor indications specified in the National Medicinal Products Administration (NMPA) approved drug instructions within 2 weeks before the first drug use;
  4. Prior treatment with anti-angiogenic therapy, immune checkpoint inhibitor therapy, or any treatment targeting immune costimulatory factors, which target the immune mechanism of tumor immune action;
  5. Patients who received immunoregulatory drugs within 2 weeks before the first dose;
  6. Non-resolved toxicity of grade 1 or higher than Common Terminology Criteria for Adverse Events (CTCAE) due to any previous treatment, excluding alopecia, peripheral sensory impairment.
* Comorbidities and medical history:

  a. Decompensated cirrhosis and active hepatitis; b. Kidney abnormalities: i. Renal failure requiring hemodialysis or peritoneal dialysis; ii. Presence of clinically significant hydronephrosis that, in the judgment of the investigator, cannot be resolved by nephrostomy or ureteral stent placement.

  c. Cardiovascular and cerebrovascular abnormalities: i. Myocardial ischemia or myocardial infarction occurred within half a year; ≥ class 2 Congestive heart failure of New York Heart Association (NYHA); Arterial thrombotic events block ≥ Grade 2; Arrhythmias that cannot be stably controlled with drugs and those that may potentially affect the trial treatment; ii. Arterial thrombotic events / venous thrombotic events, such as cerebrovascular accident, deep vein thrombosis, and pulmonary embolism, occurred within 6 months; iii. Patients with poor blood pressure control after standard treatment; iv. Previous history of myocarditis or cardiomyopathy. d. Gastrointestinal abnormalities: i. Active or documented inflammatory bowel disease, active diverticulitis; ii. Gastrointestinal perforation, fistula, and intra-abdominal abscess occurred within 6 months before the first medication; iii. The presence of clinical manifestations of gastrointestinal obstruction or the need for routine parenteral rehydration, parenteral nutrition, or indwelling gastric tube.

  e. History of immunodeficiency: i. A history of immunodeficiency, including Human Immunodeficiency Virus (HIV) positive or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation; ii. Active autoimmune disease requiring systemic therapy occurred within 2 years before the first dose. Alternative therapies are not considered systemic treatments; iii. is diagnosed with immunodeficiency or is receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy (at a dose >10mg/ day of prednisone or other iso-efficacy hormone) and continues to use it within 2 weeks of the first dose.

  f. Risk of bleeding: i. Bleeding, clotting disease, or current use of warfarin, aspirin, or other antiplatelet drugs within 28 days before the first dose; ii. Patients with any history of bleeding or coagulopathy, regardless of severity; iii. Major surgical treatment or significant traumatic injury within 28 days prior to the first dose, or locally invasive procedure within 1 week), or elective major surgical treatment required during the study; iv. Wounds or fractures that have not healed for a long time. g. Poorly controlled diabetes: fasting blood glucose (FBG) > 10mmol/L; h. Severe active or uncontrolled infection (≥CTC AE grade 2 infection); i. People with known active syphilis and active tuberculosis; j. Previous or existing interstitial pneumonia, (non-infectious) pneumonia requiring corticosteroid therapy, or other pneumonia of grade ≥2; k. Severe hypersensitivity reaction after the use of monoclonal antibodies; l. Known to have any contraindications to cisplatin/carboplatin or paclitaxel or to be allergic to any of their components; m. Those who have a history of psychotropic drug abuse and cannot quit or have mental disorders; n. Those who suffer from epilepsy and need treatment.
* Those who participated in clinical trials of other anti-tumor drugs within 4 weeks before the first drug use or did not exceed 5 drug half-lives.
* History of live attenuated vaccine vaccination within 28 days before the first dose or planned live attenuated vaccine vaccination during the study period.
* According to the investigator's judgment, there are concomitant diseases that seriously endanger the safety of the subjects or affect the completion of the study, or there are other reasons that the subjects are not suitable for enrollment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Investigator-assessed objective response rate (ORR) | Baseline to CR or PR ,about 12 months
  The proportion of subjects who achieve a prespecified reduction in tumor volume and maintain the minimum time requirement, including complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Progression free survival (PFS) | Baseline up to PD or death, about 24 months
  The time between the first dose of medication and disease progression (PD) or death before PD; If there was no PD or death before PD, the date of the last imaging assessment was used as the cutoff date.
Disease control rate (DCR) | Baseline up to PD or death, about 24 months
  The proportion of patients whose tumors shrink or remain stable for a certain period of time, including CR, PR, and stable disease (SD) cases.
Duration of response (DOR) | Baseline up to PD or death, about 24 months
  It refers to the time between the first assessment of the tumor as CR or PR to PD or death before PD in subjects with CR or PR; If subjects with CR or PR did not present with PD or die before PD, the date of the last imaging assessment was used as the cutoff date.
Overall survival (OS) | Baseline up to die, about 36 months
  The time from the first treatment to death from any cause.
PFS rate (≥6 months) | Baseline up to PD or death, about 24 months
  The proportion of patients alive and free of disease progression from the beginning of the first treatment to 6 months.
Adverse event rate | Baseline to the end of the study, about 2 years
  Occurrence of all adverse events (AEs), serious adverse events (SAEs), treatment-related adverse events (TEAEs), and immune-related adverse events (IRaes).
European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-C30 (QLQ -C30) | Baseline to the end of the study, about 2 years
  For questions 1 to 28, choose a number from 1 to 4, where 1 means no and 4 means very good. For questions 29 and 30, choose a number from 1 to 7, where 1 means very poor and 7 means very good.
European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ -CX24) | Baseline to the end of the study, about 2 years
  EORTC QLQ-CX24 is a questionnaire for measuring the quality of life of patients with cervical cancer. It has 24 items, including 3 multi-dimensional dimensions of symptoms, body image and sexual/vaginal function, and 6 single-dimensional dimensions of sexual activity, sexual enjoyment, sexual anxiety, lymphedema, menopausal symptoms and peripheral neuropathy. "None" to "very" were scored from 1 to 4, and the score was inversely proportional to the quality of life.
EuroQol 5 Dimensions (EQ-5D) Health questionnaire | Baseline to the end of the study, about 2 years
  EQ-5D is a simple health measure developed by the European Society for Quality of Life. The EQ-5D mainly consists of two parts: the EQ-5D description system and the EQ-5D Visual Analogue Scale (EQ-VAS). The EQ-5D description system describes the health status in five dimensions: mobility, self-care, daily activities, pain/discomfort, and anxiety/depression. The EQ-VAS is to record the self-rated health status of the respondents. The scale is 0-100, with 0 being "worst imagined health" and 100 being "best imagined health."
PD-L1 and TGF-β expression | At baseline
  PD-1/TGF-β double antibody can increase Leukocyte differentiation antigen 8 (CD8+) T cells in the tumor, reduce immunosuppressive myeloid cells, and inhibit PD-1/PD-L1 pathway on the basis of targeting and neutralizing TGF-β in the tumor microenvironment, which can restore the activity of T cells, enhance the immune response, and more effectively improve the inhibition of tumor.
Human papillomavirus (HPV) expression | At baseline
  The relationship between human papillomavirus and cervical cancer is very close. Persistent infection of high-risk human papillomavirus is one of the high risk factors for cervical cancer.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian